CLINICAL TRIAL: NCT05479916
Title: The Impact of Milk Protein Glycation on Protein Digestion and Absorption in Healthy Young Men
Brief Title: The Impact of Milk Protein Glycation on Protein Digestion and Absorption
Acronym: VerLys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: METC 22-004
Record Dates: First submitted 2022-07-14; First posted 2022-07-29 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Protein Digestion & Absorption
Keywords: Protein digestion; Protein glycation; Processing

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, cross-over intervention study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomized, double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low glycated milk protein (Experimental): 40 grams of low glycated milk protein, blocked lysine level ~5%
  Interventions: Dietary Supplement: Low glycated milk protein
- High glycated milk protein (Experimental): 40 grams of high glycated milk protein, blocked lysine level ~50%
  Interventions: Dietary Supplement: High glycated milk protein

INTERVENTIONS:
Dietary Supplement: Low glycated milk protein — 40 grams of protein dissolved in 600 mL of water
  Arms: Low glycated milk protein
Dietary Supplement: High glycated milk protein — 40 grams of protein dissolved in 600 mL of water
  Arms: High glycated milk protein

SUMMARY:
Rationale: Protein intake is an essential stimulus for muscle protein anabolism. The muscle protein synthetic response to protein ingestion is mainly determined by the post-prandial plasma amino acid response. Milk protein often undergoes glycation during commonly applied milk processing procedures (Maillard reaction). We have previously shown that glycated protein results in lower postprandial amino acid levels. The level of protein glycation in processed dairy products might therefore be an important modulator of the overall protein quality of a product, and its ability to stimulate protein metabolism. However, it has not yet been investigated if the glycation level of dietary protein modulates its appearance in plasma as amino acids.

Objective: To compare the appearance of dietary protein-derived amino acids in plasma after ingestion of a milk protein powder with different levels of protein glycation in healthy young men.

Study design: Double blinded, randomized cross-over study. Study population: 15 healthy young males, aged 18-35 years. Intervention (if applicable): All subjects will perform two experiments in a double-blinded, randomized order: ingest 40 g of milk protein with 5% glycation level in 600 mL water, or 40 g of milk protein with 50% glycation level in 600 mL water. After ingestion, blood samples will be taken at regular intervals during a 6 hour period.

Main study parameters/endpoints: The primary endpoint will be the appearance of milk protein-derived amino acids in plasma over the full assessment period (6 h), as determined using stable isotope tracer methodology.

DETAILED DESCRIPTION:
Proteins are mainly required as building blocks for muscle maintenance and muscle growth. To supply these building blocks for growth and development, proteins need to be well digested, and absorbed in the circulation.

Processing of milk to produce dairy products, such as milk protein powders, may affect protein quality. Heat processes can impact native protein structure, for example by inducing protein denaturation and aggregation. In addition, reducing sugars such as lactose can react with the amino group of amino acids, known as the Maillard reaction or protein glycation. Glycation levels in milk protein powders can range from 5-50%, depending on factors such as water content and storage temperature.

Several in vitro and animal studies have shown that protein glycation decreases protein digestibility. In addition, we have recently demonstrated that protein glycation reduces post-prandial amino acid availability in humans. This reduced postprandial amino acid availability could mostly be attributed to a reduction in postprandial availability of the essential amino acid lysine. The lower post-prandial availability of amino acids following ingestion of protein with a high glycation level suggests an impaired digestion and absorption of glycated dietary protein.

Therefore, to test whether ingestion of a high glycated milk protein results in a lower appearance of dietary protein-derived amino acids, a human trial has been designed. Subjects will consume a low or high glycated milk protein drink, where after several blood samples will be taken to assess the appearance of dietary protein-derived amino acids over time by using a continuous amino acid tracer infusion. The low and high glycated protein drinks reflect the lower and upper range of protein glycation reported in dairy protein products. We hypothesize that protein glycation attenuates the appearance of dietary protein-derived amino acids in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged between 18-35 years
* Healthy, recreationally active (participating in recreational sports activities ≥ 1 and ≤ 6 h per week, with a maximum of 2 h resistance-type exercise)
* 18.5 ≤ BMI ≤ 30 kg/m2
* No physical limitations (i.e. able to perform all activities associated with daily living in an independent manner).

Exclusion Criteria:

* Smoking
* Lactose intolerant or allergies to milk proteins
* Musculoskeletal disorders
* Metabolic disorders
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescribed acne medications).
* Chronic use of gastric acid suppressing medication or anti-coagulants
* Unstable weight over the last three months
* Diagnosed GI tract disorders or diseases
* Blood donation in the past 2 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Plasma appearance of dietary amino acids | 0-6 hours
  Appearance of milk protein-derived amino acids in plasma over the full assessment period (6 h), as determined using stable isotope tracer methodology

SECONDARY OUTCOMES:
Whole-body protein kinetics | 0-6 hours
  total rate of appearance, exogenous rate of appearance, endogenous rate of appearance, rate of disappearance
Whole body protein metabolism | 0-6 hours
  Protein synthesis, breakdown, oxidation, and net balance
Peak plasma lysine concentration | 0-6 hours
  Maximum plasma lysine concentration
Overall plasma amino acid responses | 0-6 hours
  Plasma amino acid concentration before and after intake of the drink
Plasma glucose concentrations | 0-6 hours
  Plasma glucose concentrations
Plasma insulin concentrations | 0-6 hours
  Plasma insulin concentrations

OTHER OUTCOMES:
Age | Baseline
  Age in years
Body weight | Baseline
  Body weight in kg
Body length | Baseline
  Body length in cm
BMI | Baseline
  BMI in kg/m^2, calculated from weight and length
Fat mass | Baseline
  Fat mass in kg.
Fat percentage | Baseline
  Fat mass in fat percentage, calculated using fat mass & body weight in kg.
Lean body mass | Baseline
  Lean body mass in kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Lieshout GA, Trommelen J, Nyakayiru J, van Kranenburg J, Senden JM, Gijsen AP, Verdijk LB, Pellikaan WF, Bragt MC, van Loon LJ. Protein glycation compromises the bioavailability of milk protein-derived lysine in vivo in healthy adult males: a double-blind, randomized cross-over trial. Am J Clin Nutr. 2025 Apr;121(4):804-815. doi: 10.1016/j.ajcnut.2025.01.025. Epub 2025 Jan 25. PMID 39870248